CLINICAL TRIAL: NCT05788159
Title: An Open Label, Balanced, Randomized, Two-Treatment, Two-Period, Two-Sequence, Two-way Crossover, Oralcomparative Pharmacokinetic（PK）Study of Lacosamide Extended-Release Tablets , Adult, Human Subjects Under Fasting Conditions.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Overseas Pharmaceuticals, Ltd. (Industry)
Collaborators: Beijing Capton Pharmaceutical Technology Development Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CS3156
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Lacosamide
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Intervention Model Description: Test preparation (T): Lacosamide extended release tablets Specification: 100mg/tablet Lot number: 22121301 Content: 100mg/tablet Expiration date: December 12, 2024 Storage conditions: Store at 20℃~25℃, short-term can be at 15C~30℃ Manufacturer: Overseas Pharmaceutical,Ltd.
  Reference preparation (R): Lacosamide Tablets Specification: 50mg/tablet Lot No.: 7883201 Content: 50mg/tablet Expiration date: September 2026 Storage condition: not more than 30C in airtight storage Manufacturer: Aesica Pharmaceuticals GmbH
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lacosamide extended release tablets (Experimental): Test preparation (T): Lacosamide extended release tablets Specification: 100mg/tablet Lot number: 22121301 Content: 100mg/tablet Expiration date: December 12, 2024 Storage conditions: Store at 20℃~25℃, short-term can be at 15C~30℃ Manufacturer: Overseas Pharmaceutical,Ltd.
  Interventions: Drug: Lacosamide Tablets
- Lacosamide Tablets (Active Comparator): Reference preparation (R): Lacosamide Tablets Specification: 50mg/tablet Lot No.: 7883201 Content: 50mg/tablet Expiration date: September 2026 Storage condition: not more than 30C in airtight storage Manufacturer: Aesica Pharmaceuticals GmbH
  Interventions: Drug: Lacosamide extended release tablets

INTERVENTIONS:
Drug: Lacosamide Tablets — Reference preparation (R): Lacosamide Tablets Specification: 50mg/tablet Lot No.: 7883201 Content: 50mg/tablet Expiration date: September 2026 Storage condition: not more than 30C in airtight storage Manufacturer: Aesica Pharmaceuticals GmbH
  Arms: Lacosamide extended release tablets
Drug: Lacosamide extended release tablets — Test preparation (T): Lacosamide extended release tablets Specification: 100mg/tablet Lot number: 22121301 Content: 100mg/tablet Expiration date: December 12, 2024 Storage conditions: Store at 20℃~25℃, short-term can be at 15C~30℃ Manufacturer: Overseas Pharmaceutical,Ltd.
  Arms: Lacosamide Tablets

SUMMARY:
An Open Label, Balanced, Randomized, Two-Treatment, Two-Period, Two-Sequence, Two-way Crossover, Oralcomparative Pharmacokinetic（PK）Study of Lacosamide Extended-Release Tablets , Adult, Human Subjects Under Fasting Conditions.

Main purpose:

To the Overseas Pharmaceutical,Ltd. Developed lacoxamide slow-release tablets (specification: 100mg) for the test preparation, UCB produced rasoxamide tablets (trade name: VIMPAT®, specification: 50mg) for the reference preparation, compare the fasting state of oral test preparation and reference preparation in Chinese healthy subjects blood concentration and main pharmacokinetic parameters, to evaluate the biological equivalence of test preparation and reference preparation.

Secondary objective:

To evaluate the safety of the test sustained-release tablets and reference tablets in the healthy Chinese subjects.

DETAILED DESCRIPTION:
A single-center, randomized, open, two-cycle, double-crossover, fasting trial design method was used. All subjects were required to sign an informed consent form prior to participation in the trial. Physical screening was performed from day -7 to day -1 of dosing, and 24 healthy subjects (containing both male and female subjects with appropriate gender ratio) who passed the screening were randomly divided into 2 groups, T-R group and R-T group, with 12 subjects in each group. The enrolled subjects were admitted to the phase I ward of the clinical research center 1 day before each cycle of dosing and fasted for more than 10 h before each cycle of dosing.

On the morning of the dosing day, after the blank blood sample collection was completed, group T received 1 tablet (100mg/tablet, Overseas Pharmaceutical,Ltd.) of lacosamide extended-release tablets developed by Overseas Pharmaceutical,Ltd. orally; group R received 1 tablet (50mg/tablet, VIMPAT®, UCB) of lacosamide orally while administering 240ml of warm water, and again 12 hours later Lacosamide 1 tablet (50mg/tablet, VIMPAT®, UCB). Standard lunch was consumed 4h after the first dose and standard dinner was consumed 10h later. No water (except 240ml of water for dosing) was allowed before and 1h after dosing, and a uniform diet was required during the trial. The second cycle was conducted in the same way as the first cycle of the test, with an elution period of 7 days.

PK blood collection and blood sample handling. For the test preparation. Before (0h) and 0.25h, 0.50h, 1.00h, 1.50h, 2.00h, 4.00h, 5.00h, 6.00h, 7.00h, 8.00h, 10.00h, 12.00h, 14.00h, 16.00h, 18.00h, 20.00h, 24.00h, 36.00h, 48.00h, 60.00h, and 72.00h for a total of 21 time points for elbow venous blood collection.

For the reference formulation. Blood was collected at 0.25h, 0.50h, 1.00h, 1.50h, 2.00h, 3.00h, 4.00h, 6.00h, 8.00h, 12.00h, 12.50h, 13.00h, 13.50h, 14.00h, 15.00h, 16.00h, 18.00h, 20.00h, 24.00h, 36.00h and 72.00h before (0h) and after dosing. 24.00h, 36.00h, 48.00h, 60.00h, and 72.00h. A total of 23 time points of elbow venous blood was collected, 4.0 ml of blood was drawn (blood collection tubes were pre-labeled with a 4 ml scale), placed in labeled EDTA-2K anticoagulation tubes, and immediately after blood collection, the blood collection tubes were gently and completely inverted three times and mixed with anticoagulant and immediately placed in an ice-water bath at 4°C for After the centrifugation operation, the samples were removed from the centrifuge and the plasma was taken from the crushed ice surface and promptly dispensed into the corresponding labeled EP tubes in 2 tubes (test tube and backup tube), both the test tube and the backup tube were no less than 500 μL. The plasma was temporarily frozen in the -20℃ refrigerator and transferred to the -80℃ refrigerator for storage after the 72h blood collection.

Vital signs (including temperature, pulse and blood pressure) were measured in the sitting position 1 hour before and 2±0.5h, 8.0h±0.5h, 24±0.5h and 48±0.5h after dosing. Physical examination, vital signs, electrocardiogram and laboratory tests were performed when the subjects were ready to leave the group after the last dose of blood was collected. Subjects were observed and asked about their subjective perceptions and possible adverse reactions and events during the course of the study. All subjects will be followed up 10 days after the end of the last dose and asked if any subsequent adverse events occurred and if AE occurred, the AE should be recorded and followed up. If an AE occurs during the trial, follow-up until the end of the AE is required.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged 18 to 60 years old (including 18 and 60 years old) with appropriate sex ratio.
2. Body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females; body mass index (BMI) within the range of 19~26.0 kg/m2 (including the critical value).

   BMI = weight (kg)/[height (m)]2.
3. Good health status, no abnormalities with clinical manifestations in the respiratory, circulatory, digestive, urinary, hematological, endocrine, immune, neurological, or psychiatric systems.
4. Subjects (including partners) have no plans to become pregnant and voluntarily use appropriate contraception from 2 weeks prior to screening until 6 months after the end of the study.
5. Subjects who are able to communicate well with the investigator and who understand and comply with the requirements of this study. Subjects who fully understand the purpose, nature, methods, and possible adverse effects of the trial, volunteer to be a subject, and sign an informed consent form prior to the start of any study procedures.

Exclusion Criteria:

1. Persons with a history of allergy to the study drug or its excipients (e.g. lactose), or allergy to drugs, food, pollen or with a history of specific allergies (asthma, allergic rhinitis, eczema), etc.
2. Those who have special dietary requirements and cannot accept a uniform diet
3. those with a history of dysphagia or any gastrointestinal disorder that affects drug absorption
4. those who cannot tolerate venipuncture and those who suffer from needle sickness and blood dizziness
5. clinically significant hematological, endocrine, cardiovascular, hepatic, renal, or pulmonary diseases that may affect drug absorption, distribution, metabolism, or excretion
6. history of surgical procedures or having taken study drugs or participated in other drug clinical trials within 3 months prior to the study
7. blood donation or significant blood loss (>450 ml) within 3 months prior to the study
8. who have taken a special diet (including dragon fruit or grapefruit and products containing grapefruit ingredients) or had strenuous exercise or other factors affecting the absorption, distribution, metabolism, or excretion of the drug within 7 days prior to taking the study drug
9. have taken any prescription medication (including birth control pills) within 14 days prior to the administration of the study drug
10. have taken any over-the-counter medication, herbal or nutraceutical product (except contraceptives) within 14 days prior to taking the study drug
11. regular drinkers of alcohol within 6 months prior to the study, i.e. more than 14 units of alcohol per week (1 unit = 360 ml of beer or 45 ml of spirits at 40% alcohol or 150 ml of wine)
12. Those who smoked more than 5 cigarettes per day in the 3 months prior to the study and did not pass the nicotine screen.
13. ingested chocolate, any caffeine-containing, or xanthine-rich food or beverage such as coffee, strong tea, cola, etc. 48 hours prior to taking study medication
14. Those who have consumed any alcohol-containing product or screened positive for alcohol within 48 hours prior to taking the study drug
15. Female subjects who have a positive pregnancy test or are breastfeeding during the screening period or during the trial
16. positive for hepatitis B surface antigen, positive for hepatitis C antibody, positive for HIV antibody or positive for primary syphilis screening
17. Those who screen positive for drugs or have a history of drug abuse within the past five years or have used drugs in the three months prior to the test
18. Subjects with an underlying medical, psychiatric, psychological or other inappropriate condition, poor compliance, or who, in the opinion of the investigator, are unsuitable for participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from time zero to the time of the last quantifiable plasma concentration of the period (AUC0-last) | Time Frame: 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation) of AUC0-last within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Area under the curve from time zero to infinity (AUC0-inf) | Time Frame: 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of AUC0-inf within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Peak concentration at each treatment period (Cmax,tp) | Time Frame: 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of Cmax,tp within [0.8, 1.25] range will be used to determine the result of bioequivalence.

SECONDARY OUTCOMES:
Peak concentration of the first dosing (Cmax) | Time Frame: 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Time to reach peak concentration of the first dosing (Tmax) | Time Frame: 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Terminal half-life (T1/2) | Time Frame: 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Mean residence time (MRT) | Time Frame: 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China